CLINICAL TRIAL: NCT00737841
Title: Effect of Bifidobacterium on Irritable Bowel Syndrome
Acronym: PBIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tohoku University (Other)
Responsible Party: Shin Fukudo, Tohoku University Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Probio-Bifid-IBS
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: stress; brain-gut interactions; visceral perception; gastrointestinal motility; emotion
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Bifidobacterium breve
  Interventions: Drug: Bifidobacterium breve
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bifidobacterium breve — 1.0 g of Bifidobacterium breve, taking orally, 3 times a day for 8 weeks.
  Arms: A
Drug: Placebo — 1.0 g of placebo, taking orally, 3 times a day for 8 weeks.
  Arms: B

SUMMARY:
There has been no data on effect of Bifidobacterium breve on symptoms of patients with irritable bowel syndrome (IBS). We hypothesized that Bifidobacterium breve is effective on symptoms of IBS patients.

DETAILED DESCRIPTION:
There has been no data on effect of Bifidobacterium breve on symptoms of patients with irritable bowel syndrome (IBS). We hypothesized that Bifidobacterium breve is effective on symptoms of IBS patients. IBS patients will be enrolled via advertisement. Any IBS subtypes will not be rejected. They will take either 1.0 g of Bifidobacterium breve 3 times a day or same amount of placebo for 8 weeks. IBS symptoms and allied markers will be checked before, during, and after the administration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBS with Rome II definition

Exclusion Criteria:

* Diagnosis of serious diseases (both physically and mentally)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-08 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Adequate relief and SIBSQ | 2, 0, 2, 4, 8 weeks during treatment and 4 weeks after treatment

SECONDARY OUTCOMES:
Psychometric test, bowel gas, blood, and feces. | 2, 0, 2, 4, 8 weeks during treatment and 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shin Fukudo, MD, PhD, Principal Investigator — Tohoku University
Locations (1):
- Tohoku University Graduate School of Medicine, Sendai, Miyagi, Japan